CLINICAL TRIAL: NCT07230470
Title: Comparative Study of Working With the LoKomat® Exoskeleton VS C-Mill® Treadmill for Gait Recovery in Rehabilitation and Improvement of Quality of Life in Adult Stroke Patients. Randomised Clinical Trial.
Brief Title: Comparative Study of LoKomat® Exoskeleton VS C-Mill® Treadmill for Gait Recovery in Rehabilitation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia de Salamanca (Other)
Responsible Party: Principal Investigator, Jorge Velazquez, PhD. Physiotherapy, Universidad Pontificia de Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06/05/2025; NCT06970314 (obsolete NCT alias)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke; Quality of life; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lokomat (Experimental): To compare the effectiveness of gait rehabilitation work in adult stroke patients using the Lokomat® tool vs.
  stroke with the Lokomat® tool.
  Interventions: Device: Lokomat®
- C-Mill (Active Comparator): Exoelectric walking aid for patients who have suffered a stroke
  Interventions: Device: C-Mill

INTERVENTIONS:
Device: Lokomat® — To compare the effectiveness of gait rehabilitation work in adult stroke patients using the Lokomat® tool vs.
  stroke with the C-Mill® tool
  Arms: Lokomat
Device: C-Mill — Exoelectric walking aid for patients who have suffered a stroke
  Arms: C-Mill

SUMMARY:
The use of robotic technology for the treatment of gait in neurological pathologies has provided different results in scientific evidence. In patients with some types of acquired brain damage, such as stroke, the use of Lokomat® therapy can bring improvements in aspects such as gait speed and balance, among other parameters and report greater functional recovery in subacute patients with greater deterioration. Similarly, the use of another technological element such as the C-Mill® reports improvements in various aspects of ambulation and balance in gait treatments for stroke patients. Likewise, the impact on the person's recovery is not only beneficial for gait rehabilitation, but also improves the perception of well-being, which can be positive in the process of readaptation to daily life.

The effect of both treatments for gait rehabilitation in adults with stroke and their impact on quality of life in the neurorehabilitation clinic will be studied.

adults with stroke and their impact on quality of life at the Lescer neurorehabilitation clinic Lescer, Madrid (Spain). Participants will be assessed at baseline, 4 weeks, 8 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke (haemorrhagic and/or ischaemic) by a specialist physician. .
* Subjects who are cognitively capable and who sign the informed consent form.

Exclusion Criteria:

* Severe cognitive impairment (Mini-Mental State Examination < 24.), or impairment that prevents correct understanding of the correct understanding of the messages and explanatory orders of the treatment and its conditions.
* Diagnosis of concomitant neurological diseases and craniocerebral trauma. cranioencephalic trauma.
* Other diseases that interfere with the gait process (e.g. disabling arthritis or arthrosis, other neurological diseases, other neurological diseases).

disabling arthritis or osteoarthritis, other concomitant neurological diseases, etc.).

- Contraindications of the robotic tools themselves.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
quality of life scale | 12 weeks
  QoL39 scale. 0 minimum - 100 maximum (higher scores mean a better outcome).
Spasticity index | 12 weeks
  Tardieu scale 0 min - 5 max (higher scores mean a worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lefeber N, De Keersmaecker E, Henderix S, Michielsen M, Kerckhofs E, Swinnen E. Physiological Responses and Perceived Exertion During Robot-Assisted and Body Weight-Supported Gait After Stroke. Neurorehabil Neural Repair. 2018 Dec;32(12):1043-1054. doi: 10.1177/1545968318810810. Epub 2018 Nov 12. PMID 30417724
- [Result] Celedova L, Krsiak M, Janku I. Immunomodulator adamantylamide dipeptide antagonizes benzodiazepine-induced rota-rod deficit in mice. Act Nerv Super (Praha). 1989 Dec;31(4):291-3. No abstract available. PMID 2638119
- [Result] Park J, Kim TH. The effects of balance and gait function on quality of life of stroke patients. NeuroRehabilitation. 2019;44(1):37-41. doi: 10.3233/NRE-182467. PMID 30741699
- [Result] Callaly EL, Ni Chroinin D, Hannon N, Sheehan O, Marnane M, Merwick A, Kelly LA, Horgan G, Williams E, Harris D, Williams D, Moore A, Dolan E, Murphy S, Kelly PJ, Duggan J, Kyne L. Falls and fractures 2 years after acute stroke: the North Dublin Population Stroke Study. Age Ageing. 2015 Sep;44(5):882-6. doi: 10.1093/ageing/afv093. Epub 2015 Aug 12. PMID 26271048